CLINICAL TRIAL: NCT05301621
Title: Accelerometry in Follow up of Arthritis - a Pilot Study
Acronym: WIAp
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helse Forde (Other)
Responsible Party: Principal Investigator, Pawel Mielnik, Consultant in Rheumatology, Helse Forde
Other Study IDs: 249395
Record Dates: First submitted 2022-03-19; First posted 2022-03-31 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Arthritis, Rheumatoid; Spondyloarthritis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arthritis patients: It is not planned any intervention. The patients' group will be invited to 4 visits.
  Interventions: Other: Akcelerometry follow up
- Healthy controls: No intervention planned. Only one visit will be conducted.
  Interventions: Other: Akcelerometry follow up

INTERVENTIONS:
Other: Akcelerometry follow up — The patients and control group will be followed up with single accelerometer.

SUMMARY:
This is a proof-of-concept study. The main goal is to evaluate if the accelerometry signal recorded from patients with arthritis in different disease activity stages, allows for assessment of the activity status. It will also be analysed if the accelerometry signal can be classified as registered in arthritis patients vs. registered in healthy control. Arthritis subjects will be recruited from the outpatients' clinic of the Rheumatology Department Helse Førde, Førde, Norway. Healthy control subjects will be recruited from the same administrative area as the patients and will be invited to participate via announcement on the Helse Forde Medical Trust website. Four visits to the site are planned for the arthritis group and one for the control group. The patients will be recruited in the active phase of arthritis as defined in the inclusion criteria.

The study's secondary objective is to develop methods for analysing the accelerometry signal in arthritis patients.

DETAILED DESCRIPTION:
Study type: Observational, proof-of-concept

Objectives:

Primary objective: To evaluate if an accelerometer signal in patients with active arthritis differs from the signal taken in inactive arthritis and healthy individuals.

Secondary goals:

* To evaluate how the accelerometer signal differs depending on the disease activity status
* To elaborate the methods for analysing accelerometry in the arthritis patients
* To build knowledge and data for future studies
* To evaluate software and hardware used

Subjects and methods:

Subjects will be recruited two groups:

1. Patient with one of the following conditions: rheumatoid arthritis, psoriatic arthritis or spondyloarthritis. All subjects must satisfy inclusion/exclusion criteria.
2. Healthy individuals as defined in inclusion/exclusion criteria

The arthritis patients with active disease will be included from the outpatients clinic of the Rheumatology Department Helse Førde Medical Trust. The healthy controls will be recruited via announcement on the Helse Førde website. The maximum number of participants is estimated for 50 subjects per group.

There will be four visits in the arthritis group and a single visit in the control group.

Following data will be collected:

For both groups: age, gender, anthropometric data (high, weight, limbs length), information about comorbidities and used drugs.

Additionally, from arthritis patients disease activity data will be collected: tender joint count, swollen joint count, overall patients/physician assessment, MHAQ, BASDAI, CRP and ESR.

At all visits, ball participants will perform a set of simple physical activities such as walking, clapping, arm swinging, and moving small subjects on the table. The accelerometry signal will be recorded during those exercises.

Study management:

An interim analysis is planned after data is collected from the first 5-10 participants. The steering committee will assess study progress at this stage and decide about further study conduct.

ELIGIBILITY:
Inclusion Criteria:

Patients:

1. Clinical diagnosis of rheumatoid arthritis (RA), psoriatic arthritis (PsA) or spondyloarthritis (SPA).
2. Planned or newly started (within 4 weeks before baseline visit) disease-modifying treatment.
3. Disis activity defined as:

   * RA - DAS28 (ESR or CRP) minimum 3.2,
   * PsA - DAPSA minimum 15,
   * SPA - BASDAI minimum 4.0.
4. A minimum number of tender or swollen joints:

   * RA - 4/4,
   * PsA - 2/2,
   * SPA - not applicable.
5. Subject without comorbidities defined in the exclusion criteria.
6. Willing to participate and consent competent.
7. Over 18 years old.

Controls:

1. Without any inflammatory rheumatic disease
2. Without any comorbidity as defined in the exclusion criteria.
3. Willing to participate and consent competent.
4. Over 18 years old.

Exclusion Criteria:

Both patients and controls:

1. Chronic neurologic disorders such as multiple sclerosis, parkinsonism, active epilepsy, symptomatic peripheral neuropathy, sequels after radiculopathy or other central nervous system deficit.
2. Paresis after cerebral stroke (mild deficits or TIA can be allowed).
3. Serious heart failure (NYHA 3 or above).
4. Pregnancy.
5. Active psychotic disorder.
6. Activ alcohol or drug addiction.
7. Fast use of medicine that can significantly influence CNS function (low dose sleeping medicine 12 hours before a visit can be allowed).
8. Spinal compression fractures less than six months before baseline.
9. Other limb fractures, within 4 months before baseline if it can influence patient's mobility
10. Other medical conditions that can influence patient's mobility

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be collected from Rheumatologic outpatients clinic Helse Forde. Only patients with the active disease will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of arthritis activity status | 2023
  Analysis of raw akcelerometry will be used to detect disease activity status

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Mielnik, MD, PhD, Principal Investigator — Helse Forde
Locations (1):
- Pawel Mielnik, Førde, Vestlandet, Norway

IPD SHARING:
Plan to Share IPD: No